CLINICAL TRIAL: NCT01032850
Title: Sorafenib in Combination With Capecitabine for Patients With Measurable Hepatocellular Carcinoma
Brief Title: Sorafenib With Capecitabine for Patients With Measurable Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0820; NCI-2011-02945 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Results first posted 2015-07-17 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2016-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: INST 0820; sorafenib; capecitabine; hepatocellular carcinoma; lung; nexavar; xeloda; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Sorafenib & Capecitabine (Experimental): Intervention: Sorafenib & Capecitabine: Sorafenib twice a day by mouth (400mg) Capecitabine twice a day by mouth (850mg)
  Interventions: Drug: Sorafenib & Capecitabine

INTERVENTIONS:
Drug: Sorafenib & Capecitabine — Intervention: Sorafenib twice a day by mouth (400mg), Capecitabine twice a day by mouth (850mg). One cycle of treatment will consist of capecitabine on days 1-7 and 15-22 while sorafenib will be given daily continuously. Cycles will be repeated every 28 days.
  Other Names: Sorafenib; Capecitabine; Nexavar; Xeloda

SUMMARY:
This research study will evaluate Sorafenib (Nexavar®) and Capecitabine (Xeloda®) to see the following:

* how effective this combination of study drugs will be in treating HCC
* how long subjects respond to these study drugs
* what types of side effects can be expected, and
* how severe the side effects are

All subjects in this study will receive:

* Sorafenib twice a day by mouth
* Capecitabine twice a day by mouth

Treatment will be given in a 28-day treatment cycle.

Subjects will take sorafenib every day of the cycle. Subjects will take capecitabine on days 1-7 and 15-21 of the cycle

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC), also known as primary liver cancer, is the most common form of liver cancer and is responsible for 80 percent of the primary malignant liver tumors in adults. It is the fifth most common cancer in the world. HCC disproportionately affects men, with four times as many men developing the disease as women. In 2002, approximately 626,000 cases of HCC were reported worldwide (15,000 in the United States and 53,600 in Europe), and more than 600,000 deaths (about 13,000 Americans and 57,000 Europeans) due to HCC were reported. The five-year relative survival rate is about seven percent.

The Gem-Ox regimen has been used in the treatment of pancreatic cancer with encouraging results. Preliminary results of the Gem-Ox combination have been encouraging as well.Based on these observations the possibility of adding bevacizumab, a monoclonal antibody against VEGF, is being studied by other investigators. However, the combination of GEM-OX with bevacizumab is unlikely to be tolerated by HCC patients with Child-Pugh class B and C liver cirrhosis especially those with significant thrombocytopenia.It would seem therefore that the agents that could be tolerated by cirrhotic patients with advanced HCC would include capecitabine, erlotinib and sorafenib. We propose this phase II trial of sorafenib + capecitabine combination in patients with HCC and advanced liver cirrhosis who have a platelet count of ≥ 40,000 and a Child-Pugh (C-P) class A-and B liver cirrhosis with a life expectancy of ≥16 weeks.

ELIGIBILITY:
Inclusion Criteria:

Histologic diagnosis of hepatocellular carcinoma The lesion or lesions are not resectable with curative intent. Prior loco-regional treatment (resection, RFA, chemoembolization) is allowed.

Adequate bone marrow function:

* Absolute neutrophil count (AGC) >1500/µL
* Platelet count >60,000 /µL

Renal function:

* Serum creatinine < 2.0 mg/dl, and a calculated CCT of > 30 mL/min. Hepatic function:(Patients with a Child-Pugh (C-P) class A-B)
* Bilirubin < 2.8 mg/dl (provided the Child-Pugh class of liver cirrhosis is A or B (7) (ie. The Child-Pugh score is only 7 points)
* ALT and AST ≤ 5.0 times the ULN • Hemoglobin > 8.5 g/dl

ECOG/Zubrod/SWOG Performance Status = 0>1 Life expectancy > 16 weeks Male or female' age >18 years Patients of childbearing potential must be using an effective means of contraception.

INR < 1.5 or a PT/PTT within normal limits.

Exclusion Criteria:

* Any prior systemic therapy including chemotherapy of targeted agents
* Uncontrolled ascites defined as not easily controlled by stable doses of diuretics.
* Pregnant or lactating females
* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Uncontrolled' clinically significant dysrhythmia
* History of prior malignancy within the prior 3 years, with the exception of non-melanoma carcinomas of the skin, carcinoma in situ of the cervix or breast, Rai Stage I chronic lymphocytic leukemia and superficial bladder cancer.
* Prior radiotherapy to an indicator lesion unless there is objective evidence of tumor growth in that lesion
* Uncontrolled metastatic disease of the central nervous system
* Radiotherapy within the 2 weeks before Cycle 1' Day 1
* Surgery within the 2 weeks before Cycle 1' Day 1
* Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection.
* Patients with chronic Hepatitis B or C infections are eligible.
* Active clinically serious infection > CTCAE Grade 2.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Z. Patt, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (3):
- United States (3):
  - University of New Mexico Cancer Center @ Lovelace Medical Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Cancer Center at Presbyterian Hospital, Albuquerque, New Mexico

REFERENCES:
- [Derived] Patt Y, Rojas-Hernandez C, Fekrazad HM, Bansal P, Lee FC. Phase II Trial of Sorafenib in Combination with Capecitabine in Patients with Hepatocellular Carcinoma: INST 08-20. Oncologist. 2017 Oct;22(10):1158-e116. doi: 10.1634/theoncologist.2017-0168. Epub 2017 Jul 7. PMID 28687627
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 participants were screened. 39 did not meet criteria; 2 refused study entry. 15 participants were enrolled.
Groups:
- Arm 1: Sorafenib & Capecitabine: Intervention: Sorafenib & Capecitabine: Sorafenib twice a day by mouth (400 mg) Capecitabine twice a day by mouth (850 mg)
  Sorafenib & Capecitabine: Intervention: Sorafenib twice a day by mouth (400 mg), Capecitabine twice a day by mouth (850 mg). One cycle of treatment will consist of capecitabine on days 1-7 and 15-22 while sorafenib will be given daily continuously. Cycles will be repeated every 28 days.
Period: Overall Study
Arm/Group | Arm 1: Sorafenib & Capecitabine
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: Sorafenib & Capecitabine
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 61 [54 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: The primary objective of the study is to evaluate safety and tolerability of the study treatment regimen. The analyses will be descriptive and no formal hypotheses testing will be performed. Toxicities (i.e. Adverse Events) are evaluated prior to each treatment and during any clinical visit.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Arm 1: Sorafenib & Capecitabine
Number analyzed (Participants) | 13
participants
  Thrombocytopenia | 9
  Neutropenia | 1
  Low phosphate levels | 3
  Low magnesium levels | 2
  Low calcium levels | 2
  Low sodium levels | 1
  High bilirubin levels | 3
  Elevated aspartate aminotransferase | 2
  Hand and foot syndrome | 3
  Mucositis | 1
  Alopecia (Hair loss) | 1
  Skin rash | 1
  Deep vein thrombosis | 3
  Treatment related deaths | 0

2. Secondary Outcome: Disease Control Rate of Response (DCR)
Description: Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI:) Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Disease control rate (DCR) is the sum of the percentages of patients achieving complete and partial responses and stable disease
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Sorafenib & Capecitabine
Number analyzed (Participants) | 13
percentage of participants
  Complete Response (CR) | 8
  Partial Response (PR) | 8
  Stable Disease (SD) | 61
  Disease Control Rate of Response (DCR) | 77

3. Secondary Outcome: Overall Survival (OS)
Description: The time from treatment initiation to death by any cause
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Sorafenib & Capecitabine
Number analyzed (Participants) | 13
Months | 12.7 [8.5 to 23.4]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The time from treatment initiation to disease progression or death by any cause. Progression is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI:) Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Sorafenib & Capecitabine
Number analyzed (Participants) | 13
months | 4.15 [2.1 to 5.5]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm 1: Sorafenib & Capecitabine
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Sorafenib & Capecitabine (N=13)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hyponatremia (Low sodium levels) (Metabolism and nutrition disorders) | 1 (1)
Anorexia (lack of appetite) (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Death (General disorders) | 1 (1) — Number of treatment-related deaths
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Sorafenib & Capecitabine (N=13)
Blurred Vision (Eye disorders) | 1 (1)
Eye disorders - other (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Ascites (Accumulation of fluid in the abdomen) (Gastrointestinal disorders) | 6 (12)
Oral hemorrhage (bleeding gums) (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (18)
Dyspepsia (Heartburn) (Gastrointestinal disorders) | 3 (4)
Mucositis: oral (Mouth inflammation) (Gastrointestinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 6 (11)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (7)
Edema (General disorders) | 2 (2)
Edema: face (General disorders) | 1 (1)
Edema: limb (General disorders) | 5 (8)
Fatigue (General disorders) | 7 (17)
Flu like symptoms (General disorders) | 1 (1)
Hepatotoxicity (General disorders) | 1 (1)
Mucosal Infection (Infections and infestations) | 1 (1)
Respiratory infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Hernia surgery (Injury, poisoning and procedural complications) | 1 (1)
Hernia surgery repair (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Elevated bilirubin (Investigations) | 3 (13)
Elevated creatinine (Investigations) | 1 (1)
Hemoglobin decreased (Investigations) | 1 (6)
Hyperglycemia (Increased blood glucose) (Investigations) | 1 (1)
Hypoalbuminemia (Decreased albumin levels) (Investigations) | 4 (7)
Hypocalcemia (Decreased calcium levels) (Investigations) | 3 (5)
Hypokalemia (Decreased postassium levels) (Investigations) | 1 (1)
Hypomagnesemia (Decreased magnesium levels) (Investigations) | 2 (7)
Hyponatremia (Decreased sodium levels) (Investigations) | 6 (8)
Hypophosphatemia (Decreased phosphate levels) (Investigations) | 4 (7)
Increased Bilirubin (Investigations) | 1 (1)
Laboratory abnormality - Other (Investigations) | 1 (1)
Leukocytes decreased (Investigations) | 1 (1)
Neutrophils decreased (Investigations) | 2 (4)
Platelets decreased (Investigations) | 4 (22)
Weight loss (Metabolism and nutrition disorders) | 7 (10)
Anorexia (Loss of appetite) (Metabolism and nutrition disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain: Other (Musculoskeletal and connective tissue disorders) | 4 (9)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Paresthesia (Numbness, tingling) (Nervous system disorders) | 2 (3)
Altered mental state (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Nosebleed) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (low blood oxygen) (Reproductive system and breast disorders) | 2 (2)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Hair loss) (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Hand and foot syndrome (Skin and subcutaneous tissue disorders) | 6 (16)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritis (Itching) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hypertension (High blood pressure) (Vascular disorders) | 4 (6)
Hypotension (Low blood pressure) (Vascular disorders) | 1 (1)
Intracerebral hemorrhage (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes